CLINICAL TRIAL: NCT00376402
Title: Phase II Study of a Pandemic Influenza Vaccine in Elderly Participants
Brief Title: Study of a Pandemic Influenza Vaccine in Elderly Participants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seqirus (Industry)
Responsible Party: Dr Russell Basser, CSL Limited
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CSLCT-PAN-05-24
Record Dates: First submitted 2006-09-11; First posted 2006-09-14 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2008-11

CONDITIONS: Influenza
Keywords: Pandemic; Influenza; Prevention; Vaccine; Prevention of Pandemic Influenza
MeSH Terms: conditions — Influenza, Human

INTERVENTIONS:
Biological: H5N1 Pandemic Influenza Vaccine

SUMMARY:
The World Health Organisation has warned that an influenza pandemic is inevitable. The avian influenza H5N1 virus strain is one of the leading candidates to cause the next influenza pandemic. The elderly are likely to be a special target group for vaccination; therefore, this study will test the safety and immunogenicity of a H5N1 pandemic influenza vaccine in a healthy elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female participants

Exclusion Criteria:

* History of clinically significant medical conditions
* History of Guillain-Barre syndrome or active neurological disease
* Resident of nursing home or long-term care facility

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 200
Dates: Start 2006-10; Study Completion 2007-06

PRIMARY OUTCOMES:
Safety and immunogenicity

CONTACTS AND LOCATIONS:
Overall Officials: Peter Richmond, Dr, Principal Investigator — Princess Margaret Hospital for Children
Locations (2):
- Australia (2):
  - CMAX, a division of IDT Australia, Adelaide, South Australia
  - Princess Margaret Hospital for Children, Perth, Western Australia